CLINICAL TRIAL: NCT03320564
Title: A Study to Assess the Impact of Moderate/Significant Infiltrations on the Standardized Uptake Values of Target Lesions
Brief Title: Infiltration Effect on SUV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment slow due to improved extravasation rate.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Lucerno Dynamics, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00046320; LUC-2017-001 (Other Grant/Funding Number: Lucerno Dynamics, LLC)
Record Dates: First submitted 2017-10-19; First posted 2017-10-25 (Actual); Results first posted 2019-04-03 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2019-03

CONDITIONS: Dose Response Relationship, Drug
Keywords: injections, intravenous; fluorodeoxyglucose F-18

STUDY DESIGN:
Intervention Model Description: All patients with a moderate or greater infiltration on a routine F-18 FDG PET will be invited to return for a repeat scan.
Masking Description: Reader will not be informed which scan was infiltrated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Infiltration (Experimental): Repeat F-18 FDG PET
  Interventions: Diagnostic Test: F-18 FDG PET

INTERVENTIONS:
Diagnostic Test: F-18 FDG PET — Repeat scan performed by specially trained staff to reduce risk of repeat infiltration.

SUMMARY:
A widely used semi-quantitative parameter to assess tumor status is the standardized uptake value (SUV). SUV estimation accuracy can be impacted by many variables. Today there still exists a significant amount of variability in PET/CT results in test and re-test studies. This variability can be introduced by instrumentation and subject-specific factors. Variability reduces image quality and increases the required changes in tumor quantification to reflect real tumor response or progression.

PET/CT scanning process requires that the entire net injected dose of radiolabeled tracer is administered intravenously as a bolus. The quality and quantification of a PET/CT image is highly dependent on the uptake of radiolabeled tracer. Boellaard et al. have indicated infiltrations could potentially underestimate SUV measurements by as much as 50%. Infiltrations and obstructions are not uncommon.

Recent studies using a novel QA/QC tool (LaraTM System) for the radiotracer injection process revealed that current means to detect infiltration do not completely identify all infiltrations/obstructions. Since infiltrations may not be visible in the standard field of view (FOV) and since the impact of a peripheral circulatory obstruction may not be visible even if an injection site is in the FOV, it is possible for reading and treating physicians to be unaware that a patient's image and quantification has been impacted. Additionally, when current means do detect an infiltration, they under-represent the severity because they are not capturing that infiltrations often resolve during the uptake period. As a result, infiltrations or obstructions may cause SUV inaccuracy and could adversely impact staging and tumor assessments.

The purpose of this study will be to characterize the impact of moderate or greater infiltrations on standardized uptake values. Patients experiencing a moderate or greater infiltration on a routine clinical PET scan will be invited to return for a repeat scan with injection performed by specially trained personnel to reduce the risk of repeat infiltration. The two scans will be compared to assess for changes in tumor uptake intensity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with solid tumors undergoing PET/CT scan who have at least one measurable target lesion and sustain a moderate or greater infiltration.

Exclusion Criteria:

* Subjects unwilling or unable to tolerate a repeat PET/CT scan.
* Subjects with meaningful medical intervention between PET/CT scans that would likely impact SUV.
* Subjects with follow up injection infiltrations that would likely impact the SUV.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shane C Masters, MD, PhD, Principal Investigator — Wake Forest Baptist Health, Department of Radiology
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osman MM, Muzaffar R, Altinyay ME, Teymouri C. FDG Dose Extravasations in PET/CT: Frequency and Impact on SUV Measurements. Front Oncol. 2011 Nov 16;1:41. doi: 10.3389/fonc.2011.00041. eCollection 2011. PMID 22655246
- [Background] Silva-Rodriguez J, Aguiar P, Sanchez M, Mosquera J, Luna-Vega V, Cortes J, Garrido M, Pombar M, Ruibal A. Correction for FDG PET dose extravasations: Monte Carlo validation and quantitative evaluation of patient studies. Med Phys. 2014 May;41(5):052502. doi: 10.1118/1.4870979. PMID 24784399

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infiltration
Started | 2
Completed | 1
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Infiltration
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1
Initial Lara TAC score [Mean (Standard Deviation); unit: units on a scale] — Range of values is -infinity to infinity. Less than 0 is considered non-extravasated. Greater than 1000 is considered at least moderate extravasation Larger values indicate greater severity of extravasation.
  units on a scale | 1104 (NA) — Single participant

OUTCOME MEASURES:

1. Primary Outcome: Change in SUVpeak of Target Lesions Between Infiltrated and Non-infiltrated Scans
Description: Target lesions selected as per PERCIST criteria. These criteria require more space than allowed to explain. Reference J Nucl Med 2009; 50: 122S-150S. DOI: 10.2967/jnumed.108.057307
Time Frame: Baseline scan and follow up scan within 7 days
Population: Up to 5 target lesions measured per participant (4 for this subject) with mean and standard deviation reported below.
Measure: Mean (Standard Deviation); unit: SUV (dimensionless)
Arm/Group | Infiltration
Number analyzed (Participants) | 1
SUV (dimensionless) | 3.6 (1.4)

2. Other Pre Specified Outcome: Change in Metabolic Tumor Volume of Target Lesions Between Infiltrated and Non-infiltrated Scans
Description: Metabolic tumor volume to be measured using threshold defined in PERCIST criteria
Time Frame: 7 days
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Change in Total Lesion Glycolysis of Target Lesions Between Infiltrated and Non-infiltrated Scans
Description: Total lesion glycolysis is calculated for the same metabolic tumor volume as Outcome 2
Time Frame: 7 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Estimated Tumor Stage or Predicted Response to Therapy Between Infiltrated and Non-infiltrated Scans
Description: Response is defined per PERCIST criteria
Time Frame: 7 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All subjects assessed from enrollment to study closure. For the subject with data recorded, approximately 5 months between enrollment and study closure.
Arm/Group | Infiltration
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infiltration (N=1)
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Subject hospitalized 4 days after initial PET scan due to abdominal pain ongoing prior to enrollment, attributed to the malignancy that prompted the PET scan. Repeat scan had not yet happened at this time.

LIMITATIONS AND CAVEATS:
Early study termination due to slow subject accrual with resulting sample size too small for analysis. This was mainly due to improvement in injection techniques and lower than expected extravasation rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT03320564/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT03320564/ICF_001.pdf